CLINICAL TRIAL: NCT03935711
Title: The Prevalence of Extra Root Canals and the Root Canal Configuration in Mandibular Anterior Teeth in a Sample of Egyptian Population Using Cone Beam Computed Tomography. A Hospital-based Cross-Sectional Study
Brief Title: The Prevalence of Extra Root Canals and the Root Canal Configuration in Mandibular Anterior Teeth in a Sample of Egyptian Population Using Cone Beam Computed Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Passant Yusuf Abulabas, masters degree student, Cairo University
Other Study IDs: ORAD 7-1
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Number of Root Canals and it's Configurations in Lower Anteriors
Keywords: cbct; cbct dental; mandibular anterior teeth; canal morphology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The considerable incidence of extra root canals of anterior mandibular teeth that is usually missed due to lack of knowledge and scarce studies leading to improper endodontic treatment, Therefore, endodontists are in need of additional investigations to enhance the quality of the root canal treatment to avoid failure

DETAILED DESCRIPTION:
Settings:

The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes.

Variables:

•Prevalence of extra root canals in mandibular anterior teeth - Classification and prevalence of observed types -

Data Sources / Measurements:

* Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
* Exposure parameters of the scans will vary depending on patients' sizes (according to the manufacturer's recommendations). images with 0.2 voxel size will be reviewed.
* For proper visualization of the canals number and configuration in anterior mandibular teeth, scrolling through the three orthogonal cuts and oblique reformatted planes.
* CBCT images will be interpreted by two oral and maxillofacial radiologists (with different experiences) independently; blinded from demographic data of the patients and from the results of each other.
* Vertucci classified the canal configurations of mandibular anterior teeth into four types (Vertucci, 1974) :

Type I: Single canal is present from the pulp chamber to the apex. Type II: Two separate canal leaves the pulp chamber, but join short of the apex to form one canal.

Type III: One canal leaves the pulp chamber, but it divides into two within the body of the root, the canals merge again to exist as one canal.

Type IV: Two separate and distinct canals are present from the pulp chamber to apex.

Type V: A single canal leaves the pulp chamber but divides into 2. Type VI: 2 separate canals leave the pulp chamber, join at the midpoint, and then divide again into 2 with 2 separate apical foramina.

Type VII: 1 canal leaves the pulp chamber, divides and then rejoins within the root, and finally redivides into 2 separate canals with 2 separate apical foramina.

Type VIII: 3 separate and distinct canals begin from the pulp chamber to the root apex.

* Each radiologist will evaluate the images for presence of extra root canal with a time lag of two weeks between the two reading sessions. If present, its configuration (classification) will be registered. Any disagreement will be solved by consensus between the two observers.
* If extra root canals type II , type IV or type VI is detected, then the distance between the canal orifices will be measured using built in measuring tool in the software.
* The measurements will be carried out by one observer (PY) and will be repeated 2 weeks later for intra-observer reliability assessment. Bias No source of bias.

Study Size:

Based on the Iranian paper by Haghanifar et al., 2017, the prevalence of two root canals in mandibular anterior teeth (12.1%) Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval) a total sample size of 170 mandibular anterior tooth will be sufficient. The sample size was calculated by Epi info 7 software.

ELIGIBILITY:
Inclusion criteria:

* Scans showing the anterior teeth areas.
* The teeth had to be completely developed

Exclusion criteria:

* Teeth to be examined, endodontically treated teeth.
* Teeth with crown restorations.
* Cast metal post inside the canal
* Teeth with apical lesions.
* Carious teeth
* Scans with low quality
* Dilacerated roots
* Resorbed roots

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
the number of root canal in mandibular anterior teeth | 2019
  detection number of canals in mandibular anterior teeth through Oblique Reformatted cuts,measuring unit is categorical nominal data %
the number of root in mandibular anterior teeth | 2019
  detection number of roots in mandibular anterior teeth through Oblique Reformatted cuts,measuring unit is categorical nominal data %
the root canal configuration in mandibular anterior teeth | 2019
  the consequestial configuration of root canals through Oblique Reformatted cuts,measuring unit is categorical nominal data %

SECONDARY OUTCOMES:
prevalence of multi-root canal according to gender | 2019
  detect the prevalence according to gender, measuring unit is categorical nominal data % they are either male or female.
the distance between the root canal orifices in lower anteriors | 2019
  the distance between the root canal orifices in type II, type IV or type VI ,measuring unit Built-in measuring tool (ruler) axial cut